CLINICAL TRIAL: NCT02297477
Title: Therapeutic Efficacy of Atovaquone-proguanil and Artesunate-atovaquone-proguanil for the Treatment of Uncomplicated P. Falciparum Malaria in Areas of Multidrug Resistance in Cambodia.
Brief Title: The ASAP Study - Therapeutic Efficacy of Atovaquone-proguanil vs. Artesunate-atovaquone-proguanil in Cambodia
Acronym: ASAP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Collaborators: National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other); Naval Medical Research Center, Asia (NMRC-A) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WR2115
Record Dates: First submitted 2014-10-18; First posted 2014-11-21 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — atovaquone, proguanil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- atovaquone-proguanil (AP) (Active Comparator): A standard fixed-dose 3 day regimen of Atovaquone-proguanil (AP) for treatment of uncomplicated P. falciparum malaria.
  Interventions: Drug: atovaquone-proguanil
- artesunate-atovaquone-proguanil (ASAP) (Active Comparator): A standard fixed-dose 3 day regimen of Atovaquone-proguanil (AP) plus 3 days of artesunate (200mg per day) for treatment of uncomplicated P. falciparum malaria.
  Interventions: Drug: artesunate-atovaquone-proguanil

INTERVENTIONS:
Drug: atovaquone-proguanil — A daily fixed dose combination of 4 tablets containing atovaquone 250mg and proguanil hydrochloride 100mg (total 1000mg/400mg respectively)
  Arms: atovaquone-proguanil (AP)
Drug: artesunate-atovaquone-proguanil — A daily fixed dose combination of 4 tablets containing atovaquone 250mg and proguanil hydrochloride 100mg (total 1000mg/400mg daily respectively) in addition to 4 tablets containing 50mg artesunate (200mg daily)
  Arms: artesunate-atovaquone-proguanil (ASAP)

SUMMARY:
This is a two-arm, randomized, open label Treatment Study evaluating the therapeutic efficacy, safety, tolerability and pharmacokinetics of a three-day course of Atovaquone-Proguanil (AP) or a three-day course of Atovaquone-Proguanil combined with 3 days of Artesunate (ASAP) in patients with uncomplicated Plasmodium falciparum malaria at selected sites in Cambodia. Atovaquone-proguanil, soon to adopted as a first line antimalarial agent by the National Malaria Control Program (CNM) in Cambodia in provinces with confirmed multidrug resistance, will be given with or without artesunate (AS) as a directly observed, standard three-day fixed dose combination treatment to all volunteers enrolled. The efficacy and safety of both drug combination as well as evidence for in vivo and in vitro resistance to their components will be monitored during the treatment period. All volunteers will receive a single dose of 15mg of primaquine as recommended by WHO with the first dose of AP or ASAP to block the transmission of malaria to mosquitoes. Resistance to AP and ASAP will be assessed by a combination of clinical, pharmacologic, and parasitological parameters including genomic signatures of selection during careful weekly follow-up visits for 6 weeks. Investigators will also be able to evaluate the effects of primaquine on the sexual stages of malaria (gametocytes).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with uncomplicated P. falciparum malaria (volunteers with mixed P. falciparum and P. vivax infections may be enrolled), 18-65 years of age
2. Baseline asexual parasite density between 100-200,000 parasites/microL
3. Able to provide informed consent
4. Available and agree to follow-up for anticipated study duration including 3 day treatment course at the Medical Treatment Facility, and weekly follow-up for the 42-day period.

Exclusion Criteria:

1. Allergic reaction or medical contraindication to atovaquone, proguanil, artesunate or primaquine, to include a calculated serum creatinine clearance estimate of less than 30mL/min
2. Significant acute comorbidity requiring urgent medical intervention
3. Signs/symptoms and parasitological confirmation of severe malaria
4. Use of any anti-malarial within the past 7 days, or atovaquone-proguanil in the past 30 days
5. Use of the following concomitant medications within 7 days, which may cause or be volunteers to significant drug-drug interactions with study drug - tetracycline, metoclopramide, rifampin, rifabutin, zidovudine or etoposide.
6. Pregnant or lactating female, or female of childbearing age, up to 50 years of age, who does not agree to use an acceptable form of contraception during the study
7. Judged by the investigator to be otherwise unsuitable for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy at 42 days (with 95% confidence intervals) for AP with and without artesunate for uncomplicated P. falciparum diagnosed by positive PCR-corrected malaria microscopy. | 6 weeks

SECONDARY OUTCOMES:
Efficacy at 28 days (with 95% confidence intervals) for atovaquone-proguanil and artesunate-atovaquone-proguanil for uncomplicated P. falciparum diagnosed by positive PCR-corrected malaria microscopy. | 4 weeks
Rates of sexual stage infections at days 1, 4, week 1 and week 2 based on a combined endpoint of light microscopy and PCR analysis for detection of gametocyte maturity. | 2 weeks
Comparative rates, duration and intensity of treatment-related adverse drug events, and total adverse events in each treatment group. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lek Dysoley, MD, Principal Investigator — National Center for Parasitology, Entomology and Malaria Control; Mariusz Wojnarski, MD, Principal Investigator — Armed Forces Research Institute of Medical Sciences (AFRIMS)
Locations (1):
- Anlong Veng Referral Hospital, Anlong Veaeng, Oddar Meancheay, Cambodia